CLINICAL TRIAL: NCT04994158
Title: Myeloproliferative Neoplasms Associated SplanChnic Vein Thrombosis: Mascot Registry
Brief Title: MASCOT Registry of Patients With Myeloproliferative Neoplasms Associated Splanchnic Vein Thrombosis
Acronym: MASCOT-R
Status: Completed | Type: Observational
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mallika Sekhar, Consultant Haematologist, Royal Free Hospital NHS Foundation Trust
Other Study IDs: IRAS 261989
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Myeloproliferative Neoplasm; Splanchnic Vein Thrombosis; JAK2 V617
Keywords: registry
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Drugs, procedures — standard of care only. non interventional registry.
  Other Names: cytoreductive drugs, anticoagulation drugs

SUMMARY:
A registry of UK patients diagnosed to have splanchnic vein thrombosis and myeloproliferative neoplasm, including isolated mutation of JAK2V617f. The purpose of the registry is to understand outcomes, treatment variations and data to inform and enable future clinical trial design and facilitate regulatory approval decision-making.

DETAILED DESCRIPTION:
Splanchnic or abdominal vein thrombosis (SVT) comprises thrombosis of hepatic, portal, superior mesenteric, splenic vein in isolation or combination. It has a prevalence of 1-2% in the general population based on autopsy reports. However, 40-50% of patients with hepatic vein thrombosis and about 25-30% of patients with PVT have an underlying myeloproliferative disease that is the cause of the thrombosis. Although some data on MPN-SVT have been published from European registries, the lack of sufficient clinical and scientific data in these patients has led to variation in treatment patterns with regard to timing, choice and duration of anticoagulation, the use of cytotoxic or biologic agents and interventions with thrombolysis and stenting with TIPSS in the acute stage. Data on the patterns of treatment of these patients in U.K and their outcomes with regard to morbidity and mortality are lacking. Availability of such data in U.K. will lead to the design of good quality prospective interventional studies.

PROJECT DESIGN This registry is designed for longitudinal real-world data collection on UK patients with MPN-SVT who are managed at tertiary liver centres in U.K. A pre-defined data set, built by a committee of specialist clinicians from the Mascot registry investigators will be collected and entered into the electronic web-based database built by Dendrite Clinical Systems Ltd.

The data captured includes demographic information linked to the NHS number, which will enable linked-anonymous data accrual and analysis as well as correlation with the Systemic Anti-Cancer Therapy Data Set (SACT) via the National Cancer Registration and Analysis Service (NCRAS) and Cancer Drug Fund (CDF) database. It will also allow interrogation of the national registries for stroke (SSNAP) and cardiac surgery (NACSA) as co-morbidities involving arterial circulation are prevalent in 30% of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Myeloproliferative neoplasm (MPN, WHO 2008, WHO 2016, BCSH) and splanchnic vein thrombosis
* Isolated Jak2v617f allele and splanchnic vein thrombosis
* MPN and portal cavernoma

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MPN of any category and splanchnic vein thrombosis
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
transformation of MPN | 5 years
  transformation to Myelofibrosis or leukaemia
progression of liver disease | 5 years
  progression of liver disease
thrombosis events | 5 years
  new or recurrent or improvement of thrombosis
haemorrhage events | 5 years
  haemorrhage

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Free London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data of identifiable nature will not be shared. Post analysis data will be published.